CLINICAL TRIAL: NCT02336750
Title: A Phase III Trial Comparing Dexamethasone, Aprepitant With or Without Mirtazapine in Delayed Emesis Control and Appetite Improvement
Brief Title: Adding Mirtazapine to Dexamethasone and Aprepitant for Delayed Emesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Fudan BR2014-15 CBCSG019
Record Dates: First submitted 2015-01-03; First posted 2015-01-13 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aprepitant; Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): D1:Chemotherapy Dexamethasone:7.5mg D2-4 Aprepitant:125mg D1, 80mg D2-3 Mirtazapine:15mg D2-4
  Interventions: Drug: Aprepitant; Drug: Mirtazapine
- control group (Experimental): D1:Chemotherapy Dexamethasone:7.5mg D2-4 Aprepitant:125mg D1, 80mg D2-3
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — 125mg D1, 80mg D2-3
  Other Names: Aprepitant Capsules
Drug: Mirtazapine — 15mg D2-4
  Other Names: Mirtazapine Tablets
  Arms: treatment group

SUMMARY:
Comparing Dexamethasone, Aprepitant and Mirtazapine With Dexamethasone and Aprepitant in Delayed Emesis Control and Appetite Improvement

DETAILED DESCRIPTION:
A Phase III Trial Comparing Efficacy and Safety of Dexamethasone, Aprepitant and Mirtazapine With Dexamethasone and Aprepitant in Delayed Emesis Control and Appetite Improvement

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had delayed emesis after receiving AC regimen or regimens including cisplatin, and will subsequently accept the same chemotherapy regimens
2. Karnofsky Performance Status ≥60.
3. Life expectancy of more than 3 months.
4. Hemoglobin ≥ 90 g/L (No blood transfusion within 14 days), Absolute Neutrophil Count ≥ 1.5×10^9/L, Platelet Count ≥ 75×10^9/L, Serum Bilirubin ≤ 1.5×ULN, ALT and AST ≤ 3.0×ULN (without liver metastases), ALT and AST ≤ 5.0×ULN (with liver metastases), Serum Creatinine ≤ 1×ULN, Endogenous Creatinine Clearance>60ml/min
5. Be able to read, understand and complete the questionnaire and diary, including FLIE and Food Diary. Note: Must be able to understand written Chinese.
6. Be able to understand the study procedures and sign informed consent.
7. Meet one of the followings about contraception:

For fertile women：

1. Urine pregnancy test in screening should be negative. If urine pregnancy test is positive, the patient could be enrolled only when serum pregnancy test is negative.
2. They should agree to abstinence or use double barrier methods of contraception during the research, within at least 14 days before enrolling and one month after the last dose of study medicine.
3. If taking oral contraceptives, the patient should agree to add a barrier method of contraception during the research, within at least 14 days before enrolling and one month after the last dose of study medicine.

Unfertility is defined as anyone of the followings:

1. Natural menopausal (natural menopausal ≥6 months and the serum FSH in the Postmenopausal range, or natural menopausal ≥12 months and age >45)
2. Bilateral tubal ligation
3. 6 weeks after the bilateral oophorectomy (with or without hysterectomy )

Exclusion Criteria:

1. Treatment with any other study medicine within 4 weeks before enrollment and with unrecovered toxicities.
2. Women of reproductive age (including gestation period, lactation, a desire of pregnancy, oral contraceptives only)
3. Severe visceral disease: such as history of myocardial infarction or serious epilepsy needing medicine.
4. Mental disabilities or emotional or mental disorders.
5. Another malignancy within 5 years (except for cured basal cell carcinoma of the skin and cervical carcinoma).
6. Uncontrolled disease, such as active infections (pneumonia), diabetic ketoacidosis, gastrointestinal obstruction. And other cases which would cause bias or make patients exposed to unnecessary risks.
7. Receiving any dose of systemic glucocorticoid treatment, but local or inhaled corticosteroids is allowed.
8. Benzodiazepines or opioids treatment within 48 hours before the first day of the study, except for a single daily taking of triazolam, temazepam or midazolam.

   a)Benzodiazepines or opioids given 48 hours or longer before the first day of the study are allowed and patients can continue the medication.
9. Having vomiting, retching or nausea within 24 hours before cisplatin treatment on the first day of the study.
10. Patient will receive abdominal or pelvic radiation between a week before and 6 days after the initiation of the study.
11. Prior aprepitant treatment or hypersensitivity history to any components of the study drug.
12. Cannot swallow capsules.
13. Not eligible for the study based on the investigators.
14. Patients receiving strong inducers of CYP3A4, such as carbamazepine, dipheninum, phenobarbitone, etc..

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-12; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Delayed emesis control (no vomiting and no rescue treatment during 25-120 hours after initiation of chemotherapy) | 6 days

SECONDARY OUTCOMES:
To assess safety of treatment group and control group. (number of participants with adverse events) | 9 weeks
To assess appetite improvement after adding Mirtazapine treatment by using Food Diary. | 9 weeks
To assess complete response (CR) rate during 0-24 hours after initiation of chemotherapy, to examine differences in acute emesis control after adding Aprepitant treatment. | 24 hours
To assess complete response (CR) rate during 0-120 hours after initiation of chemotherapy. | 120 hours
no rescue antiemetic therapy in 0-24 hours, 0-120 hours and 25-120 hours after initiation of chemotherapy | 24 hours; 120 hours
time to first vomiting episode, time to first rescue antiemetic therapy and time to treatment failure (based on first vomiting episode or first rescue antiemetic therapy, whichever occurs first) | 9 weeks
To assess the impact on patients' daily life activities in both acute and delayed emesis phases after chemotherapy by using the Functional Living Index -Emesis (FLIE). | 120 hours
To assess impact of nausea and vomiting on compliance of patients receiving chemotherapy. | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Cao J, Ouyang Q, Wang S, Ragaz J, Wang X, Teng Y, Wang B, Wang Z, Zhang J, Wang L, Wu J, Shao Z, Hu X. Mirtazapine, a dopamine receptor inhibitor, as a secondary prophylactic for delayed nausea and vomiting following highly emetogenic chemotherapy: an open label, randomized, multicenter phase III trial. Invest New Drugs. 2020 Apr;38(2):507-514. doi: 10.1007/s10637-020-00903-8. Epub 2020 Feb 8. PMID 32036491